CLINICAL TRIAL: NCT00197821
Title: Evaluation of the Immunogenicity and Reactogenicity of a Pneumococcal Conjugate Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Principal Investigator, Dr. Elizabeth Miller, Consultant epidemiologist, Public Health England
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PNCA
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Streptococcus Pneumoniae
MeSH Terms: interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: pneumococcal conjugate vaccine — Pneumococcal conjugate vaccine

SUMMARY:
To compare the relative immunogenicity and reactogenicity of the existing 23 valent plain pneumococcal vaccine and a 7 valent pneumococcal conjugate vaccine in healthy UK adults aged 50-80 years, and subsequent antibody persistence and response to boosting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation in the study; ages between 50 and 80 years at recruitment

Exclusion Criteria:

* Lack of adequate comprehension of the information sheet, consent form and study nurse's explanation of the study in order to give informed consent.
* Current participation in any other clinical trial
* Any vaccination in the previous month (except influenza vaccination which can be given at any time during the study)
* Prior pneumococcal conjugate vaccine (PNC)
* 23 valent pneumococcal vaccine(PPV) in last 5 years
* Severe general or local reaction to a previous dose of PNC or PPV
* Patients currently immunocompromised as listed in UK Handbook "Immunisation Against Infectious Disease" ed 1996
* Patients who have received intravenous immunoglobulin in the previous month or who will require replacement intravenous immunoglobulin during the period of the study
* Patients in whom pneumococcal vaccination (PPV) is currently recommended as per the UK Handbook "Immunisation Against Infectious Disease"
* Deferral of vaccination if acute systemic illness or temperature >38C on day of vaccination

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | Completed by dec 2008
  ELISA based asssay for serotype specific pneumococcal responses

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MBBS FRCPath, Principal Investigator — Heath Protection Agency

REFERENCES:
- [Derived] Goldblatt D, Southern J, Andrews N, Ashton L, Burbidge P, Woodgate S, Pebody R, Miller E. The immunogenicity of 7-valent pneumococcal conjugate vaccine versus 23-valent polysaccharide vaccine in adults aged 50-80 years. Clin Infect Dis. 2009 Nov 1;49(9):1318-25. doi: 10.1086/606046. PMID 19814624
- See also: Related Info — http://www.hpa.org.uk/webw/HPAweb&Page&HPAwebAutoListName/Page/1203008863939?p=1203008863939